CLINICAL TRIAL: NCT06278805
Title: Adaptation and Validation Study of the Longer- Term Unmet Needs After Stroke Questionnaire Into Turkish
Brief Title: Adaptation and Validation of the LUNS for Use in Turkey.
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Collaborators: Ankara University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Associate Professor (Clinical), Uşak University
Other Study IDs: ayk22
Record Dates: First submitted 2023-07-21; First posted 2024-02-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Disability Physical; Quality of Life
Keywords: Stroke; Unmet need; Disability; Quality of Life; Participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Participants with chronic stroke who have more than 1 year after stroke onset and who fulfill the inclusion/exclusion criteria will be included in this single-arm study.
  Interventions: Other: The reliability and validity study of the T-LUNS

INTERVENTIONS:
Other: The reliability and validity study of the T-LUNS — To test the reliability and validity of the T-LUNS, 110 chronic stroke survivors fulfilling the inclusion / exclusion criteria at the 3 study sites will be assessed. The assessment of each patient will include recording of the demographic and clinical characteristics and administration of the T-LUNS as well as the Turkish version of the Stroke Impact Scale 3.0 (SIS). For the assessment of test-retest reliability of the T-LUNS, half of the participants (n= 55) will fill in the T-LUNS again, 2 weeks after the first administration.

SUMMARY:
According to the most up-to-date knowledge, there is no Turkish comprehensive and validated instrument to assess stroke survivors' unmet needs in the longer term. So, this study aims to translate and adapt the LUNS into Turkish and examine its psychometric properties in survivors living at home after a stroke.

Our hypothesis in this study is:

- The Turkish Longer-term Unmet Needs after Stroke Questionnaire (T-LUNS) is a valid tool for assessing the unmet needs of stroke patients in the Turkish population.

DETAILED DESCRIPTION:
Stroke is one of the top causes of mortality worldwide, and has decreased in many countries, but an increasing number of stroke survivors are living with a disability after being discharged from the hospital. Approximately 25-30% of stroke patients will remain disabled and they will be largely dependent upon their family members and caregivers for their daily living activities. According to patients' perceptions of whether they have received any or enough assistance with a particular challenge, or of whether an issue has not been addressed at all or properly, unmet needs observed by stroke survivors may be practically evaluated. Also, it is critical to identify unmet requirements of stroke survivors in order to inform the delivery of health and social care services. The available data demonstrates that post-acute and chronic stroke survivors have a wide range of unmet requirements. Based on various contextual factors such as the availability of health and social care services, the number of years after stroke, the degree of disability, and demographic parameters, each stroke survivor has, on average, two to five unmet requirements. The Longer-term Unmet Needs after Stroke (LUNS) monitoring tool, is a 22-item questionnaire developed by The Longer-Term Stroke Care (LoTS care) study team (ref1). This questionnaire concerns the need for information as well as the physical, social, and emotional consequences of stroke. According to a cross-sectional study among 850 British stroke survivors, the lower LUNS scores were consistently related to poorer (mental) health according to the Short Form 12 (SF-12) (ref1). Groeneveld et al. translated and cross-culturally adapted the LUNS into Dutch and assessed its psychometric properties in chronic stroke survivors (ref2). Also, LUNS have been translated into different languages such as Korean, Brazil, and Malawi (ref3-4).

According to the most up-to-date knowledge, there is no Turkish comprehensive and validated instrument to assess stroke survivors' unmet needs in the longer term. So, this study aims to translate and adapt the LUNS into Turkish and examine its psychometric properties in survivors living at home after a stroke.

Permission has already been received from Bradford Teaching Hospitals NHS Foundation Trust.

This study will include two stages.; The stage will include the translation and adaptaion procedure of the original English version of the LUNS instrument into Turkish (LUNS-T). The second and the final stage will include the reliability and the validity study of the LUNS-T and this step will be performed according to the guidelines of Beaton et al. for the process of cross-cultural adaptation of self-report measures (ref5). Finally, we will assess the reliability and the validity of LUNS-T.

Stage 1. Translation and adaptation of LUNS into Turkish and establishment of Turkish LUNS (T-LUNS).

This stage will include translation, synthesis, back translation, expert committee review, and pretesting of the pre-final version of T-LUNS according to the guidelines for the process of cross-cultural adaptation of self-report measures proposed by Beaton DE et.al, 2000 (ref5).

Stage 2. Reliability and validity study of the T-LUNS. To test the reliability and validity of the T-LUNS, 110 chronic stroke survivors fulfilling the inclusion/exclusion criteria at the 3 study sites will be assessed. The assessment of each patient will include recording of the demographic and clinical characteristics and administration of the T-LUNS as well as the Turkish version of the Stroke Impact Scale 3.0 (SIS). For the assessment of test-retest reliability of the T-LUNS, half of the participants (n= 55) will fill in the T-LUNS again, 2 weeks after the first administration.

Sample size: It is planned to include at least 110 participants in the study with a 5:1 ratio between the sample size and the number of items (ref6).

Statistical analysis:

Mean, standard deviation, median, interquartile range, frequency, and percentage will be used as descriptive statistics. Student's t-test for continuous variables, Mann Whitney U test for ordinal variables, chi-square test, or Fisher's exact chi-square test for categorical variables will be used for comparisons between two independent groups. Cohen's kappa coefficient will be used to analyze the degree of agreement of the test-retest agreement of the scale items.

An exploratory factor analysis (EFA) for categorical data using the weighted least square method will be used to investigate the dimensionality of the item of the questionnaire (T-LUNS). Model fit will be evaluated using the root-mean-square error of approximation (RMSEA) that accounts for model parsimony. RMSEA values <0.08 suggest adequate fit; values <0.05 indicate good fit (ref7). Items with factor loadings below 0.30 will be eliminated. A p-value less than 0.05 will be considered significant. External construct validity of the T-LUNS will be tested by the investigation of the association with the relevant domains of the Stroke Impact Scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were diagnosed with stroke
* More than 1 years after the stroke onset
* Age 18 to 70 years
* Had a physical therapy and rehabilitation after stroke
* Cognitive functions are sufficient to fill in the questionnaires in the study
* Who give consent to participate in the study

Exclusion Criteria:

* Had delirium, confusion, or other severe consciousness problems
* Suffered from uncontrolled comorbid systemic medical conditions
* Unable to follow commands because of severe cognitive impairment
* Had a serious visual disturbance
* Individuals with musculoskeletal disabilities
* Currently participating in physical therapy or another interventional study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 110 chronic stroke patients who are in the follow-up of the study centers and attend for an outpatient visit at the Department of Physical Medicine and Rehabilitation
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
The Turkish Longer-term Unmet Needs after Stroke Questionnaire (T-LUNS) | through study completion, an average of 9 months
  After translation and adaptation of the LUNS into Turkish the T-LUNS will be created. The T-LUNS will be used to identify longer-term unmet needs of stroke patients in the areas of information, services, social and emotional consequences, health problems, and related areas. The T-LUNS includes 22 statements that express a need for in- formation or advice ("I would like advice on employment after stroke"); a need for assistance or aids ("I need additional aids or adaptations inside the home"); or worries or complaints ("I am worried that I might fall [again] and this is stopping me from doing usual things"). Each item has a "yes or no" response, with the "no" option applying to either no need or fulfillment of a need. Based on Rasch and factor analysis in previous research, the original developers of the LUNS considered the scale neither suitable for the calculation of a total score nor for division into domains.
The Stroke Impact Scale 3.0 (SIS) | through study completion, an average of 9 months
  The Stroke Impact Scale (3.0) is a 59-item self-report assessment of stroke outcome used to assess Health-related quality of life (HRQoL). The Stroke Impact Scale has 8 domains: strength, hand function, mobility, physical and instrumental activities of daily living (ie, ADLs and IADLs), memory and thinking, communication, emotion, and social participation. Scores for each domain range from 0 to 100, and higher scores indicate a better HRQoL. Four of the subscales (strength, hand function, ADLs/IADLs, and mobility) can be combined into a composite physical domain. The Stroke Impact Scale also includes a question (item 50) to assess the patient's global perception of recovery. The respondent is asked to rate his or her percentage of recovery on a visual analog scale of 0 to 100, with 0 meaning no recovery and 100 meaning full recovery.Turkish version of the SIS, which was validated before, will be used (ref8)

CONTACTS AND LOCATIONS:
Overall Officials: AYSUN GENC, Assoc. Prof, Principal Investigator — Ankara University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation; AYSE A KUCUKDEVECI, Prof, Principal Investigator — Ankara University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation; AYSE YALIMAN, Prof, Principal Investigator — Istanbul University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation; ATILLA H ELHAN, Prof, Principal Investigator — Ankara University, Faculty of Medicine, Department of Biostatistics; EKIN I SEN, Assoc. Prof, Principal Investigator — Istanbul University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] LoTS care LUNS study team. Validation of the longer-term unmet needs after stroke (LUNS) monitoring tool: a multicentre study. Clin Rehabil. 2013 Nov;27(11):1020-8. doi: 10.1177/0269215513487082. Epub 2013 Jun 20. PMID 23787941
- [Background] Groeneveld IF, Arwert HJ, Goossens PH, Vliet Vlieland TPM. The Longer-term Unmet Needs after Stroke Questionnaire: Cross-Cultural Adaptation, Reliability, and Concurrent Validity in a Dutch Population. J Stroke Cerebrovasc Dis. 2018 Jan;27(1):267-275. doi: 10.1016/j.jstrokecerebrovasdis.2017.08.043. Epub 2017 Sep 28. PMID 28967592
- [Background] Wellappuli NT, Perera HSR, Kasthuriratne G, Chang T, Gunawardena NS. Adaptation and validation of the Longer-term Unmet Needs after Stroke (LUNS) monitoring tool in Sri Lanka. BMC Public Health. 2023 Sep 4;23(1):1718. doi: 10.1186/s12889-023-16636-1. PMID 37667260
- [Background] Baek S, Kim WS, Park YH, Jung YS, Chang WK, Kim G, Paik NJ. Korean Version of the Longer-Term Unmet Needs After Stroke Questionnaire. Ann Rehabil Med. 2023 Oct;47(5):367-376. doi: 10.5535/arm.23044. Epub 2023 Oct 4. PMID 37907228
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Gorusch RL. Factor Analysis. 2nd ed. Hillsdale, NJ: Lawrence Erlbaum Associates; 1983.
- [Background] Hart DL, Mioduski JE, Stratford PW. Simulated computerized adaptive tests for measuring functional status were efficient with good discriminant validity in patients with hip, knee, or foot/ankle impairments. J Clin Epidemiol. 2005 Jun;58(6):629-38. doi: 10.1016/j.jclinepi.2004.12.004. PMID 15878477
- [Background] Hantal, A. O., Dogu, B., Buyukavci, R., & Kuran, B. (2014). Stroke impact scale version 3.0: study of reliability and validity in stroke patients in the turkish population/Inme etki olcegi 3, 0: turk toplumundaki inmeli hastalarda guvenilirlik ve gecerlilik calismasi. Turkish Journal of Physical Medicine and Rehabilitation, 60(2), 106-117.
- See also: International spread of the Longer-term Unmet Needs after Stroke (LUNS) questionnaire — https://ageingstrokeresearch.org/international-spread-of-the-longer-term-unmet-needs-after-stroke-luns-questionnaire/